CLINICAL TRIAL: NCT03218072
Title: A Phase Ia, Multi-centers, Open-label, Dose-escalation Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HLX01 (a Potential Rituximab Biosimilar) in Patients With CD20-positive B-cell Lymphomas
Brief Title: A Study to Evaluate Safety, Tolerability, PK and PD of HLX01 in Patients With CD20-positive B-cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX01-NHL01
Record Dates: First submitted 2017-07-07; First posted 2017-07-14 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: B-cell Lymphomas
MeSH Terms: conditions — Lymphoma, B-Cell

ARMS (3):
- HLX01 250 mg/m2 (Experimental): HLX01 250 mg/m2 administrated intravenously
  Interventions: Drug: HLX01
- HLX01 375 mg/m2 (Experimental): HLX01 375 mg/m2 administrated intravenously
  Interventions: Drug: HLX01
- HLX01 500 mg/m2 (Experimental): HLX01 500 mg/m2 administrated intravenously
  Interventions: Drug: HLX01

INTERVENTIONS:
Drug: HLX01 — a potential rituximab biosimilar

SUMMARY:
To evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of HLX01 (a potential rituximab biosimilar) in patients with CD20-positive B-cell lymphomas.

DETAILED DESCRIPTION:
This was a phase Ia, multicenter, open-label, dose-escalation clinical study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics characteristics of HLX01 injection in patients with CD20-positive B-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ aged ≤ 65 years, male or female;
* having histologically confirmed diagnosis of relapsed/refractory CD20-positive B-cell lymphomas which needed consolidation therapy;
* Eastern Cooperative Oncology Group (ECOG) performance status≤1 and life expectancy ≥3 months;
* providing signed and dated informed consents.

Exclusion Criteria:

* Usage of rituximab or other anti-CD20 monoclonal antibody within 2 years before enrollment;
* usage of hematopoietic cytokines within 1 week before enrollment, e.g. granulocyte colony stimulating factor (G-CSF);
* recent major surgery (excluding diagnostic surgery) within the past 8 weeks;
* peripheral nervous system diseases or central nervous system diseases;
* inadequate hematologic function met any of the following at screening: white blood cell count <3.0×109/L, absolute neutrophil count (lobocyte and rhabdocyte) <1.5×109/L, platelet count <100×109/L, hemoglobin <90 g/L, for patients with bone marrow involvement, absolute neutrophil count (lobocyte and rhabdocyte) <1.0×109/L, platelet count <75×109/L, hemoglobin <80 g/L;
* inadequate liver function met any of the following at screening: total bilirubin>1.5×the upper limit of normal range (ULN), ALT or AST>2.0×ULN, alkaline phosphatase (ALP)>3.0×ULN;
* abnormal renal function (serum creatinine>1.5×ULN);
* abnormal thyroid function (TSH< lower limit of normal or > upper limit of normal with clinical significance judged by investigators);
* positive test result(s) for serum HIV antigen or antibody;
* seropositivity of HBsAg, or seropositivity of HBcAb and HBV DNA>ULN; seropositivity of Anti HCV antibody;
* history of herpes zoster and left with sequelae or latent infection;
* other serious disease which may restrict subjects to participate in the trial (such as ongoing active infection, uncontrolled diabetes mellitus, severe cardiac insufficiency or angina pectoris, gastric ulcer, active autoimmune disease, etc.);
* pregnancy or breast feeding female, or not willing to use effective contraceptive measures during the study;
* allergic constitution, or known allergic to components of rituximab or other anti-CD20 monoclonal antibody;
* history of alcoholism or drug abuse; participation in other clinical trials within 3 months before enrollment;
* not suitable for enrollment at investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05-04 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
AEs | From First infusion to Day 90
  The type, severity and incidence of adverse events
SAEs | From First infusion to Day 90
  Thetype, severity and incidence of SAEs

SECONDARY OUTCOMES:
AUC0-inf | From First administration to Day 90
  Area under the serum concentration-time curve from time 0 extrapolated to infinity
Cmax | From First administration to Day 90
  Maximum serum concentration
t1/2 | From First administration to Day 90
  terminal half-life
CD19 positive B cells | From First administration to Day 90
  The count of CD19 positive in peripheral blood
CD20 positive B cells | From First administration to Day 90
  The count of CD20 positive in peripheral blood
Antidrug antibodies of HLX01 | From First administration to Day 90
  The concentration of anti-HLX01 in serum

REFERENCES:
- [Result] Shi Y, Zhang Q, Han X, Qin Y, Ke X, Su H, Liu L, Fu J, Jin J, Feng J, Hong X, Zhang X, Wu D, Jiang B, Dong X. Phase 1 studies comparing safety, tolerability, pharmacokinetics and pharmacodynamics of HLX01 (a rituximab biosimilar) to reference rituximab in Chinese patients with CD20-positive B-cell lymphoma. Chin J Cancer Res. 2021 Jun 30;33(3):405-416. doi: 10.21147/j.issn.1000-9604.2021.03.11. PMID 34321836